CLINICAL TRIAL: NCT02326402
Title: THEME Registry: TandemHeart Experiences and MEthods (THEME Registry)
Brief Title: TandemHeart Experiences and MEthods (THEME Registry)
Acronym: THEME
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: CardiacAssist, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: THEME
Record Dates: First submitted 2014-12-15; First posted 2014-12-29 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Heart Diseases; Lung Diseases
Keywords: Circulatory support; Extracorporeal circulatory support; Extracorporeal bypass; LifeSPARC
MeSH Terms: conditions — Heart Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: TandemHeart or LifeSPARC System — Percutaneous insertion of TandemHeart or LifeSPARC System
  Other Names: TandemHeart; LifeSPARC System

SUMMARY:
This study is intended to be a multicenter, prospective observation registry. By collecting prospective descriptive data, provide insight into disease defining characteristics resulting in the clinical decision to use TandemHeart® or LifeSPARC™ System for mechanical support and enhance knowledge of best practice regarding clinical management, weaning and removal/exit strategies.

DETAILED DESCRIPTION:
The TandemHeart or LifeSPARC percutaneous extracorporeal life support system is used to support circulation. The percutaneous cannulas facilitate access to the venous and arterial circulatory vessels. When connected to the TandemHeart or LifeSPARC centrifugal pump, mechanical support is provided with sufficient cardiac power to perfuse the organs of the body.

It is anticipated that THEME Registry™ analysis will provide insight into disease defining characteristics resulting in the clinical decision to use the TandemHeart or LifeSPARC System for mechanical support and enhance knowledge of best practice regarding clinical management, weaning and removal. The progression of the illness prior to, during and following support will be collected. The THEME Registry will collect descriptive data regarding patient selection criteria and the clinical management of the patient including strategies used to wean and remove the device. Specifically the objectives of the THEME Registry are:

* Summarize the characteristics of the patients who receive the System for temporary percutaneous mechanical support with or without an oxygenator, including demographics, pre-implant medical history, details of present illness, exit strategy.
* Evaluate the timing of initiation of System support in relation to the progression of the presenting illness and the association of this with clinical outcomes.
* Collect descriptive data related to clinical management of the patient while on mechanical support, including procedural details, duration of support, anticoagulation, hemodynamics and biochemical parameters to define trends in clinical care and the association of this decision-making with clinical outcomes.
* Collect hospital discharge information including Intensive Care Unit (ICU) and Hospital length of stay (LOS).
* Collect survival and exit strategy status at 30 and 180 days post-initial System insertion.
* Collect serious adverse events from the time of Pump insertion through removal of the System (or Pump).
* Provide data regarding patient characteristics and outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has had the TandemHeart or LifeSPARC System inserted percutaneously (e.g. in the cath lab or peri-operatively)
2. Age >= 18
3. Patient (or legally authorized representative [LAR]) has signed informed consent

Exclusion Criteria:

1. Patient is incarcerated (prisoner)
2. Participation in a clinical trial of an investigational drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in whom the System has been inserted percutaneously (e.g. in the cath lab or peri-operatively) for any diagnosis/condition at an institution participating in the THEME Registry (or transferred to an institution participating in the THEME Registry following insertion).
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Survival to Pump removal with myocardial and/or pulmonary recovery, durable ventricular assist device (VAD) implant or transition to another mechanical support device, or cardiac and/or lung transplant | 180 Days
  Survival

SECONDARY OUTCOMES:
Occurrence of Serious Adverse Events (SAEs) related to the device while on support | Approximately 72 hours after start of support
  Serious Adverse Events

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Princeton-Baptist Medical Center, Birmingham, Alabama
  - Banner - University Medical Center Tucson, Tucson, Arizona
  - University of California, San Diego, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - St. John's Hospital, Springfield, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. Louis University Hospital, St Louis, Missouri
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
  - Providence Sacred Heart Medical Center & Children's Hospital, Spokane, Washington
  - Medical College of Wisconsin-Froedtert Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Rao P, Mosier J, Malo J, Dotson V, Mogan C, Smith R, Keller R, Slepian M, Khalpey Z. Peripheral VA-ECMO with direct biventricular decompression for refractory cardiogenic shock. Perfusion. 2018 Sep;33(6):493-495. doi: 10.1177/0267659118761558. Epub 2018 Feb 21. PMID 29466925